CLINICAL TRIAL: NCT05148013
Title: PNF Versus Pilates Exercises on Pain, Body Image, Fear-Avoidance Beliefs, Core Stability, Disability and Balance Functions in Patients With CLBP: A Randomized Controlled Study
Brief Title: PNF vs Pilates Exercises in Patients With CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gözde İyigün, Faculty member, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/60-18
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain
Keywords: CLBP; Pilates exercise; Proprioceptive Neuromuscular Facilitation; Pyschological functions; Physical functions
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise group (Experimental): Pilates exercise group will receive a total of 20 sessions of 30 minute Pilates exercises 5 days a week which will be performed under the supervision of a physiotherapist.
  Interventions: Other: Pilates exercise
- PNF exercise group (Experimental): A total of 20 sessions of PNF exercises for 30 minutes, 5 days a week, will be performed individually with a physiotherapist.
  Interventions: Other: PNF exercise

INTERVENTIONS:
Other: Pilates exercise — All participants will be given a basic introduction to the Pilates-based exercises and will be taught how to activate the core muscles, which entails isometric contraction of the transverses abdominis, pelvic floor, and multifidus muscles while exhaling during diaphragmatic breathing, before beginning the exercise program. The Pilates exercise program will consist of floor exercises on a mat, including the following exercises: one-leg kick, single leg stretch, shoulder bridge, the hundred, one leg circle, and swimming. All exercises progressed at three degrees of difficulty: basic, intermediate, and advanced. Depending on the patient's tolerance, each exercise will be done for 8-10 repetitions. The treatment plan included a five-minute warm-up, twenty minutes of exercise, and a five-minute cool-down.
  Arms: Pilates exercise group
Other: PNF exercise — The PNF techniques utilized in the PNF exercise group will include a combination of isotonics, rhythmic stabilization, and repeated stretch. The exercises which will be performed are; (1) Trunk rotation in sitting position (1a) Chopping to the left and right and (1b) Lifting to the left and right, (2) Rolling activity (2a) Resistance to pelvic anterior patterns 2(b) Resistance to posterior patterns, 2(c) Combination of scapula and pelvis, 2(d) Combination of scapula and pelvis (i.e. asymmetrical exercise for trunk extension: the scapula moves in posterior elevation, the pelvis in posterior depression) and (3) Bridging activity (3a) Stabilize the pelvis in its neutral position, 3(b) Bridging lower trunk rotation and, 3(c) Bridging on two legs in the supine position.
  Arms: PNF exercise group

SUMMARY:
Low back pain (LBP) is a common health problem that affects people all over the world and is a leading cause of disability, affecting work performance and overall health. In patients with low back pain, spinal movements are restricted, endurance decreases, flexor, and extensor muscle strength weaken, and aerobic capacity is impaired. Exercise is an essential component in the therapy of many musculoskeletal issues and chronic disorders. In the literature, studies using Pilates exercises and PNF exercises in patients with CLBP have demonstrated that both treatments have some beneficial effects in terms of reducing pain and disability, as well as improving the functional level and quality of life. Studies in the literature showed that both methods are among the treatment methods frequently used in the clinic, but it is difficult to provide sufficient information about which method is more effective. Therefore, the aim of this study is to examine the effects of PNF and Pilates exercises on pain, body image, fear-avoidance beliefs, core stability, disability, and balance functions in individuals with CLBP.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common health problem that affects people all over the world and is a leading cause of disability, affecting work performance and overall health. Chronic LBP (CLBP) is defined as a problem that develops due to mechanical or non-mechanical causes and is characterized by pain, movement, and antalgic posture in the gluteal region and spine, limiting physical activity. In patients with low back pain, spinal movements are restricted, endurance decreases, flexor, and extensor muscle strength weaken, and aerobic capacity is impaired. It has been found that in patients with CLBP, pain creates fear of movement and avoidance belief, leading to inadequacy in physical functionality and a decrease in quality of life. Exercise is an essential component in the therapy of many musculoskeletal issues and chronic disorders. Exercise therapy addresses aims such as pain relief, relaxing, strengthening weak muscles, extending shortened muscles, minimizing mechanical stress on spinal structures, correcting posture, enhancing endurance, and quickly returning to work.

The Pilates Method is a mind-body approach to therapeutic exercises that promotes movement stability and control. Pilates focuses on body posture alignment, which includes proper head, shoulder, and pelvic girdle adjustment in a neutral position while preserving spine curvatures, as well as the axial position of the lower limbs and symmetrical weight-bearing of the feet in standing position. Back pain inhibits various motions of the lumbar spine and pelvis, and this condition weakens the stabilizer muscles, which can lead to CLBP. In the rehabilitation of patients with back pain, the stabilizer muscles are emphasized in order to decrease pain and improve muscular endurance and strength. The Pilates method utilizes principles of various accepted rehabilitation methods that have scientific support for LBP, including core strengthening. This is important since core weakness has been increasingly recognized as a biomechanical deficit in patients with LBP. The systematic review study by Wells et al (2014) indicates that Pilates exercise results in statistically significant improvements in pain and functional ability in the short term compared to usual care and physical activity in people with CLBP. Another recent systematic review by Barros et al. (2020), on the other hand, shows that the Pilates exercise program in moderate-to-high quality RCTs for the treatment of lower back pain is still insufficient.

Proprioceptive neuromuscular facilitation (PNF) is based on facilitating the responses of neuromuscular mechanisms by stimulating proprioceptors which aim to increase muscle strength, improve active movement ability, increase muscle endurance, and improve stabilization at the point where the technique is applied within the movement pattern. A systematic review and meta-analysis by Tong et al. (2014), identified that compared to controls, patients with low back pain have poorer lumbar proprioception. Furthermore, Meier et al. (2019) stated that back pain-induced disturbed or diminished proprioceptive signaling likely plays a key role in causing long-term alterations in the top-down regulation of the motor system via motor and sensory cortex remodeling. Individuals with chronic LBP showed lower acuity for detecting changes in trunk position and demonstrated significantly higher trunk repositioning errors during flexion of the back compared with pain-free individuals. Nijs et al. (2012), suggested that the presence of increased proprioceptive prediction errors might originate from reduced/disrupted proprioceptive input, probably triggered by nociceptive input. Therefore, the underlying physiological mechanisms of the PNF techniques such as autogenic inhibition, reciprocal inhibition, stress relaxation, and the gate control theory may influence the competition between the proprioceptive and nociceptive inputs, resulting in pain reduction and improved joint control. Furthermore, it has been found that PNF training can increase trunk muscular flexibility, strength, and endurance, providing support for the application of PNF training in functional improvement. Pourahmadi et al. (2020) stated in their systematic review and meta-analysis study that there was a low quality of evidence and a weak level of recommendation that PNF training had good benefits on back pain and disability in LBP patients and suggested further high-quality randomized clinical trials regarding long-term effects of PNF training.

In the literature, studies using Pilates exercises and PNF exercises in patients with CLBP have demonstrated that both treatments have some beneficial effects in terms of reducing pain and disability, as well as improving the functional level and quality of life. Studies in the literature showed that both methods are among the treatment methods frequently used in the clinic, but it is difficult to provide sufficient information about which method is more effective. Therefore, the aim of this study is to examine the effects of PNF and Pilates exercises on pain, body image, fear-avoidance beliefs, core stability, disability, and balance functions in individuals with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 30-65
* Complained of CLBP for more than 3 months without any neurological impairment
* Characterize their pain as >3 on the Visual Analogue Scale (VAS)
* Non-obese (BMI 30 kg/m2)

Exclusion Criteria:

* Different areas of back pain (for example, neck pain and upper back pain)
* Previous spinal surgery, structural deformities, spinal cord compression, pregnancy, severe cardiovascular or metabolic disease, and acute infection
* Who received any physiotherapy approach or exercise therapy in the previous three months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Visual Analogue Scale (VAS) will ve used to measure the pain severity. It is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values but is difficult to measure directly. On a 100 mm straight horizontal line, the participants will be asked to rate the intensity of their pain at rest and during exercise separately. The score was calculated using a ruler to measure the distance (mm) between the "no pain" anchor and the patient's mark on a 10-cm line, yielding a range of 0-100. A higher score indicates greater pain severity.

SECONDARY OUTCOMES:
Body Image Scale | 4 weeks
  Body Image Scale (BIS) was created in 1953 by Secord and Jourard. The first section of the original scale has 46 elements that encompass bodily components and their functions. The second section of the scale is about the self, and it comprises 55 items that examine various elements of self (personality, self-confidence, morality, etc.). The scale is a 40-item Likert scale (1: I like it very much, 5: I don't like it at all). The score of the scale ranges from 40 to 200. Higher ratings indicate greater dissatisfaction with body parts and functions.
Fear Avoidance Beliefs Questionnaire | 4 weeks
  The Fear Avoidance Beliefs Questionnnaire (FABQ) is a questionnaire that assesses how a person's fear-avoidance beliefs about physical activity and work may influence and contribute to his or her low back pain (i.e., the cognitive/affective components of pain distinct from specific tissue damage, injury, and nociception) and disability. The FABQ contains of 16 questions and 2 subscales: a "work" subscale composed of 7 items and a "physical activity" subscale composed of 4 items. The two subscales are scored separately. Another 5 additional items, which are not part of the scoring, complete the questionnaire. Patients rate their agreement with each statement on a 7-point Likert scale (0 = completely disagree, 6 = completely agree). The physical activities are scored between 0-24, while the questions about the work are scored between 0-42. The maximum score is 96, and a higher score suggests elevated fear-avoidance beliefs.
Trunk Stability Test | 4 weeks
  The Trunk Stability Test (TST) required subjects to sit on either a 65cm or 75cm Swiss ball with both feet on the ground. Ball size was determined by the height of the subject which allows both ankles to be in a neutral position (0° dorsiflexion) with the knees and hips in 90° of flexion. Subjects will be asked to sit upright with their arms across the chest and extend one knee. Three trials per leg will be gathered after the practice trial and the average of two trials was recorded. The deviations from the test posture, such as the plant foot moving, the arms being uncrossed, the elevated foot touching the ground, the eyes being open, and then reaching for the table was observed. The test is performed with both eyes open and closed.
Oswestry Disability Index | 4 weeks
  The Oswestry Disability Index (ODI) is to quantify disability for low back pain. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question is scored on a scale of 0-5 (0= no disability and 5= severe disability). The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage (ranges from 0-100). A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Fullerton Advanced Balance | 4 weeks
  The Fullerton Advanced Balance (FAB) Scale is a performance-based test that evaluates static and dynamic balance. It consists of 10 parameters; 1.Feet together, eyes closed, 2.Reach forward for an object, 3.Turn in a full circle, 4.Step up and over, 5.Tandem walk, 6.Stand on one leg, 7.Stand on foam, eyes closed, 8.Two-footed jump, 9.Walk with head turns, 10.Reactive postural control. In this multi-dimensional balance assessment, the lowest score is 0, and the highest score is 40. Higher scores indicate better balance ability.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Iyigun, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, North Cyprus Via Mersin 10 Turkey, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kofotolis N, Kellis E. Effects of two 4-week proprioceptive neuromuscular facilitation programs on muscle endurance, flexibility, and functional performance in women with chronic low back pain. Phys Ther. 2006 Jul;86(7):1001-12. PMID 16813479
- [Background] Valenza MC, Rodriguez-Torres J, Cabrera-Martos I, Diaz-Pelegrina A, Aguilar-Ferrandiz ME, Castellote-Caballero Y. Results of a Pilates exercise program in patients with chronic non-specific low back pain: a randomized controlled trial. Clin Rehabil. 2017 Jun;31(6):753-760. doi: 10.1177/0269215516651978. Epub 2016 Jun 3. PMID 27260764
- [Background] da Luz MA Jr, Costa LO, Fuhro FF, Manzoni AC, Oliveira NT, Cabral CM. Effectiveness of mat Pilates or equipment-based Pilates exercises in patients with chronic nonspecific low back pain: a randomized controlled trial. Phys Ther. 2014 May;94(5):623-31. doi: 10.2522/ptj.20130277. Epub 2014 Jan 16. PMID 24435105
- [Background] Kofotolis N, Kellis E, Vlachopoulos SP, Gouitas I, Theodorakis Y. Effects of Pilates and trunk strengthening exercises on health-related quality of life in women with chronic low back pain. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):649-659. doi: 10.3233/BMR-160665. PMID 26922845
- [Background] Areeudomwong P, Buttagat V. Proprioceptive neuromuscular facilitation training improves pain-related and balance outcomes in working-age patients with chronic low back pain: a randomized controlled trial. Braz J Phys Ther. 2019 Sep-Oct;23(5):428-436. doi: 10.1016/j.bjpt.2018.10.005. Epub 2018 Oct 17. PMID 30361077
- [Background] Areeudomwong P, Wongrat W, Neammesri N, Thongsakul T. A randomized controlled trial on the long-term effects of proprioceptive neuromuscular facilitation training, on pain-related outcomes and back muscle activity, in patients with chronic low back pain. Musculoskeletal Care. 2017 Sep;15(3):218-229. doi: 10.1002/msc.1165. Epub 2016 Oct 28. PMID 27791345